CLINICAL TRIAL: NCT05551897
Title: An Open-Label, Fixed Sequence Study in Healthy Post Menopausal Female Subjects to Assess the Pharmacokinetics of Camizestrant (AZD9833) When Administered Alone and in Combination With Itraconazole
Brief Title: A Study to Assess the Pharmacokinetics of Camizestrant (AZD9833) When Administered Alone and in Combination With Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D8532C00003; 2022-002011-35 (EudraCT Number)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Breast Cancer; Selective Estrogen Receptor Degrader (SERD); ER-Positive, HER2- Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD9833; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive a single oral dose of Camizestrant on Day 1 of treatment period 1. Following washout period of 7 to 10 days, subjects will receive Itraconazole on Days 1, 2, and 3 of treatment period 2, and single oral dose of Camizestrant plus a dose of Itraconazole on Day 1, followed by Itraconazole alone on Day 2 and Day 3 of treatment period 3.
  Interventions: Drug: Camizestrant; Drug: Itraconazole

INTERVENTIONS:
Drug: Camizestrant — Subjects will be administered a single oral dose of Camizestrant on Day 1 of treatment period 1 and treatment period 3.
  Other Names: AZD9833
Drug: Itraconazole — Subjects will be administered Itraconazole twice a day on Day 1 and once daily on Day 2 and Day 3 of treatment period 2, and once daily on Day 1, 2 and 3 of treatment period 3.

SUMMARY:
This study will be conducted in healthy post-menopausal female subjects to assess the pharmacokinetics (PK) of Camizestrant (AZD9833) when administered alone and in combination with Itraconazole.

DETAILED DESCRIPTION:
This open-label, fixed sequence study will comprise of:

* A screening period of 28 days;
* A fixed sequence of three treatment period:

Treatment Period 1: Camizestrant only, Treatment Period 2: Itraconazole only, Treatment Period 3: Camizestrant and Itraconazole in combination.

• A Follow-up Visit at 7 to 14 days after the last Camizestrant PK sample in Period 3.

There will be a washout period of 7 to 10 days between Period 1 and Period 2. Each subject will be involved in the study for approximately 8 or 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal female subjects aged 50 to 70 years with suitable veins for cannulation or repeated venipuncture
* Subjects must be post-menopausal by fulfilling the following criterion:

  a. Post-menopausal defined as amenorrhea for at least 12 months or more without an alternative medical or surgical cause and confirmed by an FSH result of ≥ 30 IU/L.
* Have a body mass index (BMI) between 19 and 35 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Must agree to not use warfarin or phenytoin (and other coumarin-derived vitamin K antagonist anticoagulants) from screening, and for 2 weeks after last administration of the study drug.

Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the subject at risk because of participation in the study
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of clinically significant cardiovascular, chronic respiratory, neurological, or psychiatric disorder
* History of or ongoing clinically significant visual disturbances including but not limited to visual hallucinations, migraine with visual symptoms, blurred vision, frequent floaters/flashes associated with other symptoms such as dizziness
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the study drug.
* Any clinically significant abnormal findings in vital signs or 12-lead Electrocardiogram (ECG).
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and Human Immunodeficiency Virus (HIV) antibody.
* Known or suspected history of drug or alcohol abuse.
* History of significant allergy or hypersensitivity.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes and nicotine replacement products) within the 3 months prior to screening.
* Use of systemic oestrogen-containing hormone replacement therapy within 6 months prior to first dose in the study.
* Have any active indication for therapeutic anticoagulation, and/or having taken an anticoagulant within 14 days of beginning the study.
* Any of the following signs or confirmation of COVID-19 infection:

  1. Subject has a positive test for SARS-CoV-2 prior to admission.
  2. Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnoea, sore throat, fatigue) or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or at admission.
  3. Subject has been previously hospitalized with COVID-19 infection within the last 12 months.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) of Camizestrant | Day 1 to Day 4 (Period 1 and Period 3)
  To assess the effect of Itraconazole on AUCinf of Camizestrant.
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) of Camizestrant | Day 1 to Day 4 (Period 1 and Period 3)
  To assess the effect of Itraconazole on AUClast of Camizestrant.
Maximum observed plasma (peak) drug concentration (Cmax) of Camizestrant | Day 1 to Day 4 (Period 1 and Period 3)
  To assess the effect of Itraconazole on Cmax of Camizestrant.

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | From Screening (Day -28 to Day -2) up to follow-up visit (7 to 14 days after last Pharmacokinetic Sample) [approximately 9 weeks]
  Safety and tolerability of Camizestrant alone and in combination with Itraconazole will be assessed.
Number of subjects with adverse events leading to the discontinuation of study drug (DAEs) | From Day 1 (period 1) up to follow-up visit (7 to 14 days after last Pharmacokinetic Sample) [approximately 9 weeks]
  Number of subjects who discontinue the study drug due to adverse events will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home